CLINICAL TRIAL: NCT03003169
Title: Mastectomy in Ambulatory Breast Surgery
Acronym: MASTAMBU
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL OBS 01
Record Dates: First submitted 2016-12-21; First posted 2016-12-26 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Mastectomy
Keywords: surgery; breast cancer; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ambulatory surgery description
  Interventions: Other: Medical questionnaire

INTERVENTIONS:
Other: Medical questionnaire — * quality of life questionnaire (EORTC QLQ-C30 and QLQ-BR23)
  * Hospital Anxiety and Depression scale
  * satisfaction care questionnaire (IN-PATSAT32)

SUMMARY:
This is a prospective observational study, involving 550 mastectomies in Lorraine Institute of Oncology, to assess care patients management of ambulatory surgical compared to standard surgery procedure.

ELIGIBILITY:
Inclusion Criteria:

* patient managed for breast cancer surgery
* age >18 years old
* understand and comply with the requirements of the study
* patient must be affiliated to a social security system

Exclusion Criteria:

* patient managed for a concomitant reconstructive surgery
* bilateral breast surgery
* patient already included in another clinical trial with an experimental molecule
* men
* patient deprived of liberty or under supervision
* neoadjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes all the patients managed for total or partial mastectomy at the institute.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Impact of the type of hospitalization (ambulatory / conventional) according to the type of surgery (total / partial mastectomy) on quality of life 15 days after Intervention. | 15 days
  Quality of life is assessed by the EORTC QLQ-C30 questionnaire BR23

SECONDARY OUTCOMES:
Impact of type of hospitalization (ambulatory / conventional) depending on the type of surgery (total / partial mastectomy) on anxiety / depression of the patient 15 days after surgery. | 15 days
  Anxiety / depressions are assessed by the Hospital Anxiety and Depression scale
Patient satisfaction by type of hospitalization (ambulatory / conventional) for each type of surgery (total / partial mastectomy) | 15 days
  Patient satisfaction is assessed by a satisfaction care questionnaire (PATSAT 32).
Complication rate within 15 days the intervention according to the type of hospitalization (ambulatory / conventional) for each type of surgery (total / partial mastectomy) | 15 jours
  Postoperative complications will be classified according to Dindo- Clavien
Estimate the conversion rate from ambulatory surgical to conventional surgery | 15 jours

CONTACTS AND LOCATIONS:
Overall Officials: MARCHAL FREDERIC, MD, PU-PH, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hejl L, Raft J, Leufflen L, Rauch P, Buhler J, Abel-Decollogne F, Routiot T, Hotton J, Salleron J, Marchal F. Quality of life, anxiety, and postoperative complications of patients undergoing breast cancer surgery as ambulatory surgery compared to non-ambulatory surgery: A prospective non-randomized study. J Gynecol Obstet Hum Reprod. 2021 Feb;50(2):101779. doi: 10.1016/j.jogoh.2020.101779. Epub 2020 May 11. PMID 32407900